CLINICAL TRIAL: NCT05998642
Title: A Phase 2 Study of Ibrutinib Combination Therapy in Transplant Ineligible Individuals With Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: Ibrutinib Combination Therapy in Transplant Ineligible Individuals With Newly Diagnosed Primary CNS Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I244
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Non-hodgkin Lymphoma
Keywords: Central Nervous System
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Methotrexate; Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methotrexate, Ibrutinib +/- Rituximab (Experimental): Cycles 1-6, q14 days Day 1: Methotrexate + Rituximab Days 6-14: Ibrutinib daily orally
  Interventions: Drug: Methotrexate; Drug: Rituximab (where available); Drug: Ibrutinib

INTERVENTIONS:
Drug: Methotrexate — 3.5mg/m2 IV
Drug: Rituximab (where available) — 375mg/m2 / 1400mg IV or SC
Drug: Ibrutinib — Dose and schedule assigned at enrollment

SUMMARY:
This study is being done to answer the following question: Can the addition of a new drug to the usual treatment lower the chance of primary central nervous system lymphoma growing or spreading?

This study is being done to find out if this approach is better or worse than the usual approach for this type of cancer. The usual approach is defined as the care most people get for Primary Central Nervous System Lymphoma (PCNSL).

DETAILED DESCRIPTION:
If a patient decides to take part in this study, the patient will get 3 months of treatment with methotrexate and ibrutinib as well as rituximab (if rituximab is given for PCNSL in the applicable province). This will be followed by treatment with ibrutinib alone for up to 2 years of total treatment time.

After finishing study treatment, and even if patients stop treatment early, the study doctor will continue to follow the patient's condition for the rest of their life or until all study results are known (in approximately 6 years), watch for side effects and keep track of the patient's health. If there are any side effects that may be related to ibrutinib, the patient will be asked to come back to the clinic every 3 months until side effects improve. If there are no side effects from ibrutinib the patient will be asked to come back to clinic every 6 months until cancer worsens, and then every 6 months may be contacted by phone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological evidence of primary central nervous system (CNS) lymphoma (PCNSL); patients with vitreo-retinal lymphoma (NHL) or cerebrospinal fluid (CSF) positive disease are eligible providing there is CNS involvement on MRI compatible with PCNSL
* Patients must be 18 years of age or older
* Patients must be ineligible (≥65 years old or comorbidities) for high-dose chemotherapy and autologous stem cell transplantation. Patients must be considered fit, as determined by the treating physician, to receive high dose methotrexate, ibrutinib and rituximab as per protocol
* Patients must have consented to the release of a tumour block from their brain tumour, if available (see Section 12.0). The centre/pathologist must have agreed to the submission of the specimen(s).
* Presence of radiological documented disease. Patients believed to have residual disease following a complete resection, even if radiology is negative or equivocal, are eligible provided they are planned for standard of care methotrexate/rituximab.
* No prior systemic therapy other than the following situations:

  * Methotrexate +/- rituximab: Patients may have received one cycle of methotrexate with or without rituximab as standard of care therapy, but must be enrolled no longer than 4 weeks after first dose of methotrexate corticosteroids for PCNSL is permitted.
  * Use of corticosteroids (topical are permitted) on study (except for short-term treatment of infusion reactions and nausea prophylaxis) is not permitted. Patients receiving corticosteroids me be eligible, providing:
* they are receiving not more than dexamethasone 8mg/day (or equivalent)
* The corticosteroid will be tapered and completely discontinued within 7 days of starting the study protocol treatment. Patients who would require continued or concurrent treatment with systemic steroids are not eligible.
* Intrathecal therapy: Patients may have received intrathecal therapy at the time of diagnostic lumbar puncture. No washout period is needed prior to enrollment.
* Previous major surgery is permitted provided that surgery occurred at least 28 days prior to patient enrollment and that wound healing has occurred. The 28 day cut-off does not apply to surgery for PCNSL; treatment may begin following brain biopsy/resection when deemed safe by the treating investigator
* No prior radiation therapy for PCNSL is allowed
* ECOG performance status 0-2, and ECOG 3 permitted if secondary to primary CNS lymphoma and expected to reverse with treatment
* Patients must be able to swallow oral medications and have no known gastrointestinal disorders that may interfere with absorption (such as malabsorption).
* Patients must have adequate organ and marrow function measured within 7 days prior to enrollment including: Absolute neutrophils ≥ 1.0 x 10^9/L (independent of growth factor support); Platelets ≥ 75 x 10^9/L; Bilirubin ≤ 1.5 x UNL; ALT ≤ 3.0 x UNL (if AST >3 x UNL consult with CTG re: eligibility); Creatinine clearance ≥ 50 mL/min
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaire in either English or French
* Patients must be accessible for treatment and follow up. Patients enrolled on this trial must be treated and followed at the participating centre
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Patients with secondary central nervous system non-Hodgkin lymphoma (NHL).
* Patients with significant third space accumulation (pleural effusions, ascites) which cannot be adequately drained in advance of methotrexate administration
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. However, patients on active anticancer therapy for other advanced or metastatic malignancies are not eligible.
* Patients with a known hypersensitivity to the study drugs or their components
* Active, uncontrolled bacterial, fungal, or viral infection within 7 days prior to enrollment. Patients with hepatitis B serology suggestive of past infection (for example anti-HB-c positive but HBsAG and anti-HBs negative) are eligible if they are HBV DNA negative are being or will be concurrently treated with anti-viral therapy. Patients with a history of hepatitis C which has been treated and is no longer active are eligible. Patients with known human immunodeficiency virus (HIV) with CD4 count < 350 cells/microliter are ineligible. Patients who are HIV positive are eligible, provided:

  * They have received antiretroviral therapy for at least 4 weeks prior to enrollment, and the anti-viral drugs used are not known to have clinically relevant drug-drug interactions with ibrutinib AND
  * HIV viral load must be < 400 copies/ml within 16 weeks prior to enrollment AND No history of opportunistic infections within the past year
* Serious illnesses or medical conditions which would not permit the patient to be managed according to protocol
* Patients may not receive concurrent treatment with other anti-cancer therapy or investigational agents while on protocol therapy
* Patients with prior allogenic bone marrow transplant or double umbilical cord blood transplantation.
* Pregnant or breastfeeding women
* Patients requiring:

  1. Anticoagulation with warfarin or equivalent vitamin K antagonists
  2. Continued requirement for therapy with a strong CYP3A inhibitor or inducer (see trial webpage for list)
  3. Corticosteroid treatment with > 8mg of dexamethasone (or equivalent) at the time of enrollment
  4. Supplements containing fish oil or vitamin E, and grapefruit juice should be avoided
* Live attenuated vaccination administered within 30 days prior to enrollment
* Patients with clinically significant cardiac disease, including:

  * angina pectoris, symptomatic pericarditis, coronary artery bypass grafting, coronary angioplasty, or stenting, or myocardial infarction in the previous 12 months;
  * history of documented congestive heart failure (New York Heart Association functional classification III-IV) or cardiomyopathy;
  * uncontrolled hypertension (per Canadian guidelines);
  * atrial or ventricular arrhythmias; patients with controlled atrial fibrillation are eligible
* Patients with distant clinically significant cardiac history should have a LVEF ≥ 50% Baseline LVEF is not required for patients with only a cardiac history of hypertension which is now controlled.
* Patients may not receive concurrent treatment with other anti-cancer therapy or investigational agents while on protocol therapy.
* Patients with prior allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Pregnant or breastfeeding women.
* Patients requiring:

  1. Anticoagulation with warfarin or equivalent vitamin K antagonists
  2. Continued requirement for therapy with a strong CYP3A inhibitor or inducer
  3. Corticosteroid treatment with > 8mg of dexamethasone (or equivalent) at the time of enrollment
  4. Supplements containing fish oil or vitamin E, and grapefruit juice should be avoided.
* Live attenuated vaccination administered within 30 days prior to enrollment, or within 30 days prior to start date of pre-study methotrexate +/- rituximab for participants who receive one cycle before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
One year progression-free survival (PFS) | 5 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR = CR+CRu+PR) and complete response (CR) rate | 5 years
1-year event-free survival (EFS) | 5 years
2-year progression-free survival | 5 years
Overall survival (OS) | 5 years
Number and severity of adverse events | 5 years
To determine the impact on cognitive functioning of ibrutinib, methotrexate, and rituximab treatment in patients with PCNSL using FACT-Cog | 5 years
To determine the impact on health-related quality of life of ibrutinib, methotrexate, and rituximab treatment in patients with PCNSL using FACT-BR | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Larouche, Study Chair — CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Quebec City, QC Canada; Anca Prica, Study Chair — University Health Network-Princess Margaret Hospital, Toronto, ON Canada
Locations (8):
- Canada (8):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - The Research Institute of the McGill University, Montreal, Quebec
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No